CLINICAL TRIAL: NCT01368796
Title: Controlled Comparison in Canadian Seniors of Seasonal Influenza Vaccines for 2011-2012
Brief Title: Comparison of 4 Influenza Vaccines in Seniors
Acronym: PCIRNRT09
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: PHAC/CIHR Influenza Research Network (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H11-01457
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Influenza Vaccine
Keywords: Vaccine; Influenza vaccine; Adjuvanted Influenza vaccine; Intradermal Influenza vaccine; Seniors; Acceptability of vaccines; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluad vaccine; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Trivalent Influenza vaccine subunit (Active Comparator): The seasonal vaccine (Agriflu, Novartis) contains egg-derived, inactivated and detergent split versions of the 3 influenza strains (tri-valent). It is given into the muscle of the upper arm at a dose of 0.5 mL.
  Interventions: Biological: Agriflu
- Adjuvanted Tri-valent Influenza Vaccine (Active Comparator): The adjuvanted vaccine (Fluad, Novartis) is made with an immune-stimulator (MF59) that contains squalene oil microdroplets and two surfactants, Tween 80 and Span 65. It is given into the muscle of the upper arm at a dose of 0.5 mL.
  Interventions: Biological: Fluad
- Intradermal Tri-valent Influenza vaccine (Active Comparator): (Intanza 15ug, Sanofi Pasteur) is an inactivated, split-virion influenza vaccine. Strains are grown in fertilized hen's eggs, inactivated with formalin and split using Triton X-100 detergent, as for TIV. The syringe is attached to a micro-needle injection system (Beckton Dickinson) that limits the depth of injection to just under the skin. It is given into the skin over the upper arm at a dose of 0.1 mL.
  Interventions: Biological: Intanza
- Trivalent Split-virion Influenza vaccine (Active Comparator): Vaxigrip, Sanofi Pasteur is an inactivated, split-virion Influenza vaccine. The 3 influenza strains are grown on fertilized eggs, concentrated, purified in a sugar-like solution, detergent split, and inactivated by formaldehyde, then diluted in phosphate buffered salt solution. A dose of 0.5 mL is given into the muscle of the arm.
  Interventions: Biological: Vaxigrip

INTERVENTIONS:
Biological: Agriflu — 0.5mL dose IM vaccination
  Arms: Trivalent Influenza vaccine subunit
Biological: Fluad — 0.5mL dose of vaccine given IM
  Arms: Adjuvanted Tri-valent Influenza Vaccine
Biological: Intanza — 0.5mL dose vaccine given IM
  Arms: Intradermal Tri-valent Influenza vaccine
Biological: Vaxigrip — 0.5mL dose vaccine given IM
  Arms: Trivalent Split-virion Influenza vaccine

SUMMARY:
Based on information from several years of looking at Influenza vaccination doctors know that:

* Older adults suffer the worst illness and most deaths caused by Influenza illness of all age groups.
* Older adults do not seem to get as good a level of protection as younger adults after getting the usual seasonal Influenza vaccine.

Because of this information doctors wonder if one of the new seasonal Influenza vaccines is more effective or more acceptable.

This study has been designed to answer some of these questions. On this study doctors will compare 2 new vaccines against the usual seasonal influenza vaccine for protectiveness using several different testing methods (including the usual tests) and for acceptability.

DETAILED DESCRIPTION:
This study is prospective, multicenter, randomized, evaluator-blinded, controlled, parallel group study of 3 licensed seasonal influenza vaccine products conducted in seniors, with a 4th vaccine included in a substudy of cellular immune responses.

Ambulatory adults 65+ years of age, in good health or with stable health conditions, given TIV within the past 2 years, will be recruited in multiple Canadian centres. Subjects can be dwelling in the community or in centers providing minimal assisted living support. A total of 930 subjects will be enrolled.

Subjects will be centrally (electronically) randomized to receive either TIV, IDV or AIV on Day 0. Three blood samples will be collected (1 pre and 2 post vaccination) to measure HAI antibody responses to each virus strain (H1N1, H3N2 and B) in each vaccine, using standardized assays. Randomly selected subsets of sera from each study group will also be tested for neutralizing antibody and for cross-protection against drift variants of H3N2, H1N1 and B viruses. In a subset of subjects in Vancouver, randomization assignments will include TIV2 and extra blood samples will be obtained 0, 21 and 72 days post vaccination for CMI testing. Safety assessments will be conducted on Day 7, Day 21 and Day 180 following vaccination. Acceptability of each product, reflecting the frequency, severity and tolerability of adverse effects, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the subject, who can be male or female
* Subjects who the investigator believes can and will comply with the requirements of the protocol (i.e. return for follow-up visits, record safety observations and able to converse with study personnel including by personal telephone)
* Age 65 years or older at Visit 1
* Generally good health (stable chronic conditions acceptable), living independently or with minimal assistance (Clinical Frailty score 1-5) (33) and able to attend clinic appointments
* Receipt of at least one dose of TIV within the previous 2 influenza seasons, documented by written record or attested by a confident personal recollection. This refers to the trivalent seasonal vaccine, not the H1N12009 pandemic vaccine.

Exclusion Criteria:

* receipt of non-study influenza vaccine for 2011-12
* receipt of any live vaccine within 4 weeks or inactivated vaccine within one week of Visit 1 or planned administration of any non-study vaccines between Visits 1 and 2
* systemic hypersensitivity to influenza vaccine, hen's eggs or other vaccine constituent (eg neomycin sulphate, kanamycin, formalin)
* severe reaction to any previous influenza vaccine or vaccine component
* bleeding disorder, including anticoagulant therapy or thrombocytopenia, that contraindicates IM injection or blood collection (does not include daily low-dose ASA).
* incapacity to provide fully informed consent or be attentive to follow-up observations, resulting from cognitive impairment, abuse of alcohol, drug addiction
* lack of telephone access, inadequate fluency in English (or French in applicable jurisdictions), uncertain availability during the 3 week study participation period or for the 6 month follow-up visit
* immune compromise resulting from disease or immunosuppressive systemic medication use within 3 months of V1
* receipt of blood or blood product within 3 months of V1
* unstable medical condition, as indicated by a requirement for hospitalization or a substantial medication change to stabilize said condition within previous 3 months
* Clinical Frailty score of 6-7 (moderately frail or severely frail)
* history of Guillain-Barré syndrome

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 953 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
HAI response | Day 0; Day 21; Day 180
  The primary outcome measures will be the 3-week post-vaccination immune (HAI) responses to the 3 vaccine strains present in each product, assessed by the EMEA/CHMP criteria for evaluation of immune responses to influenza vaccines in persons >60 years of age.

SECONDARY OUTCOMES:
Seroprotection rates using microneutralization titres and cytokine testing | Day 0; Day 21; and Day 70
  As secondary immunologic outcomes seroprotection rates will be compared between the products using a higher titer (≥160) as threshold. Microneutralization titers will be compared among products at the 3 sampling points, using sera from 100 subjects per group. Cross-protection afforded by each vaccine against drift variants of H3N2, H1N1 and B viruses will be assessed using serum panels selected from 50 subjects in each group. Cellular immune responses elicited will be compared in subgroups of 30 subjects per vaccine in the CMI subjset.
Safety and Acceptability | Days 0-6; Day 21; Day 70; and Day 180
  Safety and acceptability of the vaccines will also be examined and compared as the safety outcomes. The primary outcome measurements will be the rates of local adverse events (pain, redness, swelling, itchiness) as rates of general adverse events are not expected to differ substantially among the products.

CONTACTS AND LOCATIONS:
Overall Officials: David W Scheifele, MD, Principal Investigator — University of Britich Columbia
Locations (8):
- Canada (8):
  - University of British Columbia, VITALiTY Research Center, Vancouver, British Columbia
  - University of Manitoba, Department of Medicine, Winnipeg, Manitoba
  - Canadian Centre for Vaccinology Dalhousie University, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - The Ottawa Hospital Research Institute, University of Ottawa, Ottawa, Ontario
  - University of Toronto, Mt Sinai Hospital, Toronto, Ontario
  - McGill University Health Center - Vaccine Study Center, Montreal, Quebec
  - Unité de Recherche en Santé Publique (CHUQ),, Québec, Quebec

REFERENCES:
- [Derived] Skowronski DM, Janjua NZ, De Serres G, Purych D, Gilca V, Scheifele DW, Dionne M, Sabaiduc S, Gardy JL, Li G, Bastien N, Petric M, Boivin G, Li Y. Cross-reactive and vaccine-induced antibody to an emerging swine-origin variant of influenza A virus subtype H3N2 (H3N2v). J Infect Dis. 2012 Dec 15;206(12):1852-61. doi: 10.1093/infdis/jis500. Epub 2012 Aug 7. PMID 22872731